CLINICAL TRIAL: NCT06529900
Title: The Effects of Technological Oral Health Management on Improving Oral Health, Eating Ability, Nutritional Status, and Physical Function of the Elderly in the Community After Wearing Removable Dentures: An Example of the Agricultural County
Brief Title: The Effects of Technological Oral Health Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Kuo Ya-Wen, Professor, Chang Gung University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 111-670
Record Dates: First submitted 2024-07-22; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Oral Health; Malnutrition; Dysphagia; Sarcopenia
Keywords: the elderly in the community; oral health; nutrition; eating ability; physical function; technological oral health management; dentures
MeSH Terms: conditions — Malnutrition; Deglutition Disorders; Sarcopenia | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Mastication Training and Texture and Diet Education (Experimental): Participants in this arm will receive oral mastication training combined with texture and diet education.
  Interventions: Behavioral: oral mastication training; Behavioral: texture and diet education
- Texture and Diet Education (Active Comparator): Participants in this arm will receive texture and diet education without the oral mastication training component.
  Interventions: Behavioral: texture and diet education

INTERVENTIONS:
Behavioral: oral mastication training — Through specific exercises and techniques aimed at enhancing masticatory function and overall oral health.
  Arms: Oral Mastication Training and Texture and Diet Education
Behavioral: texture and diet education — Teach the knowledge and techniques of softening food textures.

SUMMARY:
The goal of interventional study is to for the elderly who have poor chewing and eating ability after installing removable dentures through the intervention of oral mastication training and texture and diet education, the effects on oral health, eating ability, nutrition, and physical function changes are confirmed in Elderly individuals residing in Chiayi County who are 65 years of age or older, capable of self-care, conscious, and able to communicate in Mandarin and Taiwanese. The main question it aims to answer is:

•Are there significant benefits to oral health, eating ability, nutrition, and physical function through the intervention of oral mastication training and texture and diet education? Researchers will compare changes in oral health, eating ability, nutrition, and physical functioning results to see if oral mastication training is effective.

Participants will:

* Experimental group: oral mastication training and texture and diet education.
* Control group: only texture and diet education.
* Cases were tracked in month 1 and will be tracked again in month 6.

DETAILED DESCRIPTION:
Expected Results：

1. To establish an oral mastication training and texture and diet education program for the elderly who have poor chewing and eating ability after dentures are installed.
2. Provide teaching programs tailored to the evidence-based and individualized needs of the elderly.
3. Through the implementation of evidence-based oral mastication training and a texture and diet education program, the experimental group and the control group are expected to show variations in oral health, eating ability, nutrition, and physical function over time.

ELIGIBILITY:
Inclusion Criteria:

1. residing in Chiayi County who are 65 years of age or older
2. capable of self-care, conscious
3. able to communicate in Mandarin and Taiwanese.

Exclusion Criteria:

1. non-residents of Chiayi County
2. unable to take care of themselves or are unconscious
3. demented or mentally challenged and are unable to cooperate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Oral Frailty Index-8 | Baseline, 1 month, 6 months.
  The total score was 11 points. 0-2 points: low risk, 3 points: medium risk, and 4 points or above: high risk.
Iowa Oral Performance Instrument | Baseline, 1 month, 6 months.
  It is considered abnormal for values below the 5th percentile.
Food Intake Questionnaire | Baseline, 1 month, 6 months.
  A subject with four or more 'difficult-to-eat' responses to the 14-food group questionnaire would be classified as abnormal.
Comfort Eating Scale | Baseline, 1 month, 6 months.
  On a scale of 1 to 10, where 1 represents very good (no impact, no pain) and 10 represents very bad (impact, pain).
Mini Nutritional Assessment-Short Form | Baseline, 1 month, 6 months.
  0 - 7 points: malnourished; 8 - 11 points: at risk of malnutrition; or 12 - 14 points: well-nourished.
Study of Osteoporotic Fracture | Baseline, 1 month, 6 months.
  One component was considered to be in a pre-frailty state, while two or more components indicated frailty.
Handgrip strength | Baseline, 1 month, 6 months.
  Weak hand grip strength was defined as < 26 kg for men and < 18 kg for women.